CLINICAL TRIAL: NCT06558318
Title: The Role of Temporomandibular Joint Dysfunction on Proprioception, Pain-related Parameters, and Body Awareness
Brief Title: TMJ Dysfunction: Effects on Proprioception, Pain, and Body Awareness
Status: Completed | Type: Observational
Sponsor: Nagihan Acet (Other)
Responsible Party: Sponsor-Investigator, Nagihan Acet, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: AtılımU
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Disorder
Keywords: Joint Position Sense; Quantitative Sensory Testing; Temporal summation; Cervical proprioception
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "TMJ Dysfunction" for the group with TMJ dysfunction.: This group consists of young adults aged 18-25 who have been diagnosed with temporomandibular joint (TMJ) dysfunction. The diagnosis was determined using the Fonseca Amnestic Index, where participants with a score greater than 20 were classified into this group. The participants in this group are being analyzed for proprioception, body awareness, and pain-related parameters, including pain threshold, pain tolerance, and temporal summation.
  Interventions: Other: Assessment of temporomandibular dysfunction
- "No TMJ Dysfunction" for the group without TMJ dysfunction.: This group includes young adults aged 18-25 who do not exhibit temporomandibular joint (TMJ) dysfunction. Participants in this group have a Fonseca Amnestic Index score of 20 or lower. Similar to the TMJ dysfunction group, these participants are being evaluated for proprioception, body awareness, and pain-related parameters such as pain threshold, pain tolerance, and temporal summation.
  Interventions: Other: Assessment of temporomandibular dysfunction

INTERVENTIONS:
Other: Assessment of temporomandibular dysfunction — TMJ dysfunction will be measured using the Fonseca Amnestic Index. The Fonseca Amnestic Index is used to assess the severity of temporomandibular joint (TMJ) dysfunction. The index consists of 10 questions, with each question scored as 0, 5, or 10 points, depending on the severity of symptoms. The maximum total score is 100, where a higher score indicates a more severe level of TMJ dysfunction. Therefore, patients with higher scores on the Fonseca Amnestic Index are considered to have more significant TMJ issues. Based on Fonseca scores, two groups will be formed: those with scores over 20 will be labeled 'with TMJ dysfunction,' and the others 'without TMJ dysfunction.

SUMMARY:
The term "temporomandibular joint dysfunction" (TMJ dysfunction) refers to a range of anatomical and functional problems, with or without clinical signs and symptoms, that affect the TMJ and/or the chewing muscles. It is more frequent in women and young people ages between 20 and 40. Its frequency ranges from 28% to 88%. The term "temporomandibular joint dysfunction" (TMJ dysfunction) refers to a range of anatomical and functional problems, with or without clinical signs and symptoms, that affect the TMJ and/or the chewing muscles. It is more frequent in women and young people ages between 20 and 40. Its frequency ranges from 28% to 88%. This condition is frequently disregarded because of inadequate diagnosis . Additionally, TMJ dysfunction can particularly emerge in the early stages without the presence of pain. Due to the insidious onset of the disease, especially in the early stages, other TMJ-related factors, in addition to pain-related parameters, need to be considered.Therefore, the aim of the study is to investigate the effect of TME disorder on proprioception, body awareness, and pain-related parameters including pain threshold, pain tolerance, and temporal summation in young adults.

DETAILED DESCRIPTION:
"In the study, young adults aged 18-25 will be included, with TMJ dysfunction being measured using the Fonseca Amnestic Index. Based on Fonseca scores, two groups will be formed: those scoring over 20 will be labeled 'with TMJ dysfunction,' while the others will be classified as 'without TMJ dysfunction.' Proprioception will be assessed both through self-reports using the Fremantle Neck Awareness Questionnaire and via joint position sense measured by a CROM device. Body awareness will also be evaluated using the Body Awareness Questionnaire. Pain assessment, including pain threshold, tolerance, and temporal summation, will be conducted using a pressure algometer. The 'pain threshold' will refer to the point at which a person first feels pain, 'pain tolerance' will be the last point that a person can tolerate, and 'temporal summation' will be the pain sensation evaluated after 10 repetitions of the pain threshold.

ELIGIBILITY:
Inclusion Criteria:

*Being between 18-25 years old

Exclusion Criteria:

* History of cervical spine injuries or disorders
* Chronic pain conditions or diagnosed musculoskeletal disorders
* Previous neck or spine surgeries
* Neurological or psychiatric conditions affecting proprioception or pain perception
* Use of medications influencing pain sensitivity or proprioception
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of young adults aged 18-25, including those with temporomandibular joint (TMJ) dysfunction and asymptomatic controls without TMJ dysfunction. Participants are recruited from Atılım University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
Proprioception Assessment-1 (self-reported) | Single assessment at baseline
  Evaluation of proprioception using the Fremantle Neck Awareness Questionnaire:Self-reported proprioception will be assessed using the Fremantle Neck Awareness Questionnaire. The Fremantle Neck Awareness Questionnaire (FreNAQ) typically consists of 9 items, each rated on a Likert scale from 0 to 4. The scale ranges from 0 to 36 points. Higher scores on this scale indicate impaired neck awareness.
Proprioception assessment-2 | Single assessment at baseline.
  Evaluation of proprioception with joint position sense measurement via a CROM device: Proprioception will also be assessed with joint position sense via a CROM device. After finding the target angle in right and left rotation directions, the patient is asked to repeat the target angle with their eyes closed. The difference is recorded. Three measurements are taken, and the average is calculated.

SECONDARY OUTCOMES:
Pain-related parameters | Single assessment at baseline.
  Pain assessment, including pain threshold, tolerance, and temporal summation, will be conducted using a pressure algometer. The 'pain threshold' will be the point at which a person first feels pain, the 'pain tolerance' will be the last point that a person can tolerate, and the 'temporal summation' will be the pain sensation evaluated after 10 repetitions of the pain threshold.
Assessment of body awareness | Single assessment at baseline.
  Body awareness will be evaluated using the Body Awareness Questionnaire.The Body Awareness Questionnaire (BAQ) consists of 18 items scored on a 1-7 scale. The total score is the sum of all items, with a minimum score of 18 and a maximum score of 126. Higher scores indicate better body awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Nagihan Acet, Phd., Study Director — Atılım University; Sena Nur Begen, MSc., Principal Investigator — Atılım University
Locations (1):
- Atılım University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shen S, Ye M, Wu M, Zhou W, Xu S. MRI and DC/TMD Methods Analyze the Diagnostic Accuracy of the Change in Articular Disc of Temporomandibular Joint. Comput Math Methods Med. 2022 Feb 15;2022:1770810. doi: 10.1155/2022/1770810. eCollection 2022. PMID 35211184
- [Result] Ohrbach R, Dworkin SF. The Evolution of TMD Diagnosis: Past, Present, Future. J Dent Res. 2016 Sep;95(10):1093-101. doi: 10.1177/0022034516653922. Epub 2016 Jun 16. PMID 27313164
- [Result] Türken, R., S.K. Büyük, and Y. Yasin, Diş Hekimliği Fakültesi Öğrencilerinde Temporomandibular Eklem Rahatsızlıklarının ve Ağız Sağlığı Alışkanlıklarının Değerlendirilmesi. Acıbadem Üniversitesi Sağlık Bilimleri Dergisi, 2020(2): p. 208-213.
- [Result] Pires PF, de Castro EM, Pelai EB, de Arruda ABC, Rodrigues-Bigaton D. Analysis of the accuracy and reliability of the Short-Form Fonseca Anamnestic Index in the diagnosis of myogenous temporomandibular disorder in women. Braz J Phys Ther. 2018 Jul-Aug;22(4):276-282. doi: 10.1016/j.bjpt.2018.02.003. Epub 2018 Feb 21. PMID 29519746
- [Result] Heisler AC, Song J, Dunlop DD, Wohlfahrt A, Bingham CO III, Bolster MB, Clauw DJ, Marder W, Phillips K, Neogi T, Lee YC. Association of Pain Centralization and Patient-Reported Pain in Active Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2020 Aug;72(8):1122-1129. doi: 10.1002/acr.23994. Epub 2020 Jul 21. PMID 31162824
- [Result] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Result] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Result] Mehling WE, Gopisetty V, Daubenmier J, Price CJ, Hecht FM, Stewart A. Body awareness: construct and self-report measures. PLoS One. 2009;4(5):e5614. doi: 10.1371/journal.pone.0005614. Epub 2009 May 19. PMID 19440300
- [Result] Law EY, Chiu TT. Measurement of cervical range of motion (CROM) by electronic CROM goniometer: a test of reliability and validity. J Back Musculoskelet Rehabil. 2013;26(2):141-8. doi: 10.3233/BMR-2012-00358. PMID 23640315
- [Result] Walton DM, Macdermid JC, Nielson W, Teasell RW, Chiasson M, Brown L. Reliability, standard error, and minimum detectable change of clinical pressure pain threshold testing in people with and without acute neck pain. J Orthop Sports Phys Ther. 2011 Sep;41(9):644-50. doi: 10.2519/jospt.2011.3666. Epub 2011 Sep 1. PMID 21885906
- [Result] Karaca, S. (2017). Vücut Farkındalığı Anketinin Türkçe uyarlaması: Geçerlik ve güvenirlik çalışması (Yayınlanmamış yüksek lisans tezi). Muğla Sıtkı Koçman Üniversitesi Sağlık Bilimleri Enstitüsü, Muğla.
- [Result] Onan D, Gokmen D, Ulger O. The Fremantle Neck Awareness Questionnaire in Chronic Neck Pain Patients: Turkish Version, Validity and Reliability Study. Spine (Phila Pa 1976). 2020 Feb 1;45(3):E163-E169. doi: 10.1097/BRS.0000000000003207. PMID 31425430
- [Result] World Health Organization. Oral Health SurveysBasic Methods. 4th ed. Geneva: World Health Organization; 1997. [